CLINICAL TRIAL: NCT07368751
Title: Clinical Effects of Transcutaneous Vagus Nerve Stimulation in the Treatment of Frozen Shoulder: A Randomized Controlled Trial
Brief Title: Vagus Nerve Stimulation Effect in Frozen Shoulder Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Salam Alruz, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUC-FTR-SA-01
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; Vagus Nerve Stimulation; Exercise
MeSH Terms: conditions — Bursitis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous Vagus Nerve Stimulation (tVNS) plus exercises (Experimental): the interventional group will receive active tVNS plus exercise therapy including traditional exercises and home exercises.
  Interventions: Other: Active tVNS plus exercises
- Sham controlled tVNS plus exercises (Sham Comparator): the control group will receive Sham-controlled tVNS plus exercise therapy including traditional exercises and home exercises.
  Interventions: Other: Sham controlled tVNS plus exercises

INTERVENTIONS:
Other: Active tVNS plus exercises — This program will be performed 3 times per week for 6 weeks. Each session will include 30 minutes of tVNS. Stimulation will be delivered to the auricular branch of the vagus nerve using a non-invasive transcutaneous device. Electrodes will be placed on the tragus and concha regions of the ear. in addition to traditional exercises including mobilization, ROM exercises, stretching and strengthening exercises.
  Arms: transcutaneous Vagus Nerve Stimulation (tVNS) plus exercises
Other: Sham controlled tVNS plus exercises — This program will be performed three times per week for six weeks. In each session, 30 minutes of sham tVNS will be applied, during which the device will remain inactive, in addition to traditional exercise therapy including joint mobilization, range of motion exercises, stretching, and strengthening exercises.
  Arms: Sham controlled tVNS plus exercises

SUMMARY:
The goal of this clinical trial is to learn if the addition of transcutaneous vagus nerve stimulation (tVNS) to exercise is effective in improving pain, shoulder function, shoulder range of motion, and psychological factors in adults with frozen shoulder.

The main questions this study aims to answer are:

Does adding tVNS to exercise reduce shoulder pain ? Does adding tVNS to exercise improve shoulder function and shoulder range of motion? Does adding tVNS to exercise improve psychological factors ? Does adding tVNS to exercise improve patient satisfaction?

Researchers will compare the effect of active tVNS added to exercise with sham-controlled tVNS added to exercise to determine whether adding tVNS provides additional benefits in the management of frozen shoulder.

Participants will:

Receive active tVNS plus exercise therapy or sham-controlled tVNS plus exercise therapy.

Attend supervised rehabilitation sessions 3 times per week for 6 weeks. Perform a home exercise program as instructed by the study physiotherapist.

DETAILED DESCRIPTION:
This is a randomized, double-blind (participants and outcome assessors), sham-controlled study. Participants will be recruited from a university hospital. Volunteers diagnosed with frozen shoulder who meet the inclusion criteria and are referred by an orthopedics and traumatology specialist will be included.

The study will be conducted in accordance with the ethical principles of the Declaration of Helsinki. Participants who provide written informed consent and meet the inclusion criteria will be randomized in a 1:1 ratio to either exercise therapy combined with active transcutaneous Vagus Nerve Stimulation (tVNS) or exercise therapy combined with sham-controlled tVNS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years.
* Less than 50% range of motion compared with the contralateral shoulder in at least one movement (external rotation, abduction, flexion, or internal rotation).
* More than 25% loss of range of motion in at least two movement planes compared with the unaffected shoulder.
* Increasing limitation of glenohumeral external and internal rotation during abduction from 45° to 90°.
* Shoulder pain lasting at least 3 months during activities of daily living.

Exclusion Criteria:

* Passive joint range of motion within normal limits
* External rotation range of motion <30°
* Radiographic evidence of glenohumeral arthritis
* Presence of inflammatory joint disease
* Previous treatment related to the current shoulder complaint (physiotherapy and rehabilitation, intra-articular injection, or surgery)
* Pain intensity <3 according to the Numerical Pain Rating Scale (NPRS)
* Presence of neurological deficits, cardiac disease, neuropathic disorders, or pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Shoulder Pain and Disability Index (SPADI) at weeks 6 and 12. | Change from baseline in SPADI score at weeks 6 and 12
  The Shoulder Pain and Disability Index (SPADI) will be used to assess shoulder pain and disability levels in patients. SPADI consists of 13 items and includes two subscales: pain and disability. The pain subscale consists of 5 items while the disability subscale consists of 8 items. Both subscale scores and the total score are calculated on a 0-100 scale, with higher scores indicating greater pain and disability.
Change from baseline of Numerical Rating Pain Scale (NPRS) at week 6 and week 12 | Change from baseline in NPRS score at week 6 and week 12
  Pain intensity will be assessed using the Numerical Rating Pain Scale (NPRS). Participants will be asked to rate the intensity of their shoulder pain on a scale from 0 to 10, with higher scores indicating greater pain.

SECONDARY OUTCOMES:
Change from baseline in Quick Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH) score at week 6 and week 12 | Change from baseline in QuickDASH score at weeks 6 and 12
  QuickDASH is a patient-reported outcome measure and will be used to assess upper extremity function and symptoms. The total score ranges from 0 to 100, with higher scores indicating greater functional disability.
Change from baseline in Pain Catastrophizing Scale (PCS) score at week 6 and week 12 | Change from baseline in PCS score at weeks 6 and 12
  The Pain Catastrophizing Scale (PCS) will be used to assess rumination, magnification, and helplessness related to pain. The scale yields a total score ranging from 0 to 52, with higher scores indicating greater levels of pain catastrophizing.
change from baseline in the Glenohumeral Joint Range of Motion at week 6 and week 12 | Change from baseline in range of motion at weeks 6 and 12
  Glenohumeral joint range of motion will be assessed using a universal goniometer, a widely used and reliable method for measuring shoulder joint mobility.
Change from baseline in Pain Self-Efficacy Questionnaire (PSEQ) score at week 6 and week 12 | Change from baseline in PSEQ score at weeks 6 and 12
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item self-report questionnaire designed to assess an individual's confidence in performing activities despite pain. Total scores range from 0 to 60, with higher scores indicating greater pain-related self-efficacy.
Treatment satisfaction assessed with the Global Rating of Change (GRC) Scale at weeks 6 and 12 | At weeks 6 and 12
  GRC scale is designed to measure a patient's perceived improvement or deterioration over time to determine the effect of an intervention. A 5-point scale ranging from -2 to +2 will be used (-2 = much worse, -1 = worse, 0 = no change, +1 = better, +2 = much better).

CONTACTS AND LOCATIONS:
Overall Officials: Salam Alruz, Msc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No